CLINICAL TRIAL: NCT04283916
Title: Botulinum Toxin Injection in the Treatment of Open Abdomen
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Elisa Mäkäräinen, Principal Investigator, University of Oulu
Other Study IDs: 7/2020
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Open Abdomen; Botulinum Toxin Injection
MeSH Terms: interventions — Botulinum Toxins

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Botox injection: 30 consecutive patients will have 300 IU of botulinum toxin injected to six spots in abdominal wall to gain abdominal wall musculature relaxation.
  Interventions: Drug: Botulinum Toxins

INTERVENTIONS:
Drug: Botulinum Toxins — Botulinum toxin injection to abdominal wall

SUMMARY:
Botulinum toxin has been widely approved and utilized in the treatment of complex abdominal wall hernias. Botulinum toxin has been only randomly studied in the treatment of open abdomen.

DETAILED DESCRIPTION:
30 consecutive patients who have open abdomen for any indication, will have 300 IU botulinum toxin injected in three spots in either sides of the abdomen within 72 hours of the start of open abdomen. The hypothesis is botulinum toxin relaxes abdominal wall musculature to ensure better and faster closure of the open abdomen.

ELIGIBILITY:
Inclusion Criteria:

* Open abdomen

Exclusion Criteria:

* Previous incisional hernia in midline
* Patient is not in active treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 30 consecutive open abdomen patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2020-02-21 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Abdominal wall closure | 30 days
  Duration of open abdomen treatment

SECONDARY OUTCOMES:
Intensive care time | 30 days
  Treatment time in the intensive care unit
Hospitalization | 30 days
  Time spent in the hospital
Hernia | 2 years
  Incisional hernia incidence
Re-laparotomies | 30 days
  Number of abdominal explorations
Enterocutaneus fistula | 30 days
  Enterocutaneus fistula incidence
Abdominal wall closure success rate | 30 days
  the rate of complite abdominal wall closure

CONTACTS AND LOCATIONS:
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: Undecided